CLINICAL TRIAL: NCT06574165
Title: Relationships of Affect and Neuroinflammation With Clinical Pain in Veterans With Fibromyalgia
Acronym: RAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F4807-M; IK1RX004807-01A2 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
Keywords: Chronic Pain; Inflammation; Affect; Neuroinflammation; Fibromyalgia; Exercise
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Inflammation; Neuroinflammatory Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: 6-week structured exercise intervention. The intervention will include twice weekly, center-based, aerobic exercise consisting of continuous treadmill walking. 6-week waitlist control group including phone calls twice weekly. The participants will be offered the exercise intervention at the completion of the final study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Intensity Continuous Training (Experimental): 20 Veterans living with fibromyalgia and 20 Veterans living without fibromyalgia will undergo a 6-week structured exercise intervention. The intervention will include twice weekly, center-based, aerobic exercise consisting of continuous treadmill walking. Each center-based session will include 45 minutes of aerobic exercise in addition to balance and flexibility exercises to promote cool-down. During each exercise session, participants will also be asked to wear a heart rate monitor to measure mean pulse during exercise sessions.
  Interventions: Behavioral: Moderate Intensity Continuous Training
- Waitlist Control (No Intervention): 10 Veterans living with fibromyalgia and 10 Veterans living without fibromyalgia will undergo a 6-week waitlist control. This will include phone call check-ins on the participant's pain symptoms twice weekly. At completion of the final study visit the participants will be offered the option to participate in the exercise intervention.

INTERVENTIONS:
Behavioral: Moderate Intensity Continuous Training — 6-week structured exercise intervention. The intervention will include twice weekly, center-based, aerobic exercise consisting of continuous treadmill walking. Each center-based session will include 45 minutes of aerobic exercise in addition to balance and flexibility exercises to promote cool-down. During each exercise session, participants will also be asked to wear a heart rate monitor to measure mean pulse during exercise sessions.
  Arms: Moderate Intensity Continuous Training

SUMMARY:
Fibromyalgia (FM) is a chronic pain condition that disproportionately impacts Veterans. Individuals diagnosed with FM patients experience lower self-esteem and positive affect, as well as greater levels of depression, anxiety, negative affect, and pain catastrophizing. Among those experiencing FM, clinical and experimental pain are associated with specific dispositional trait profiles, which are indexed by levels of negative affect and positive affect. Neuroinflammation and inflammation also play a role in FM- related affect and pain. Recent studies that have highlighted neuroinflammation and inflammation as physiological mechanisms associated with changes in dysregulated affect and chronic pain. Veterans with FM can ameliorate dispositional traits-i.e., increasing positive affect and reducing negative affect-by participating in exercise. However, a gap exists regarding how to optimally engage Veterans with FM in an exercise program. Thus, to fully take advantage of all potential therapeutic benefits of exercise for FM, there is a critical need to identify those factors underlying exercise engagement for FM pain management. The purpose for this study is to 1) determine associations of dispositional trait styles, neuroinflammation, and inflammation with pain outcomes in Veterans with FM; and 2) develop and design a Veteran-informed exercise program.

DETAILED DESCRIPTION:
The investigators propose to recruit 30 Veterans with FM and 30 Veterans without FM who will undergo magnetic resonance spectroscopy imaging (MRSI) scans, pain assessments, and semi-structured interviews. The participants will undergo a 6-week moderate intensity continuous training exercise intervention and follow-up MRSI scans, pain assessments, and semi-structured interviews. The investigators central hypothesis is that dispositional trait styles, neuroinflammation, and inflammation will be associated with pain outcomes and exercise will induce beneficial anti-inflammatory changes. The research objective of this proposal is two-fold: 1) to acquire data on the associations between dispositional trait styles, neuroinflammation, inflammation, and pain in Veterans with FM and 2) to develop a Veteran-informed exercise program with potential to modify dispositional trait styles, neuroinflammation, inflammation, and pain in Veterans with FM.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Veterans living with FM:

* Inclusion Criteria (FM) Age 19 years or older
* Widespread pain index (WPI) 7 and symptom severity scale (SSS) score 5 OR WPI 4-6 and SSS score 9
* Generalized pain, defined as pain in at least 4 of 5 regions, is present
* Symptoms have been present at a similar level for at least 3 months
* A diagnosis of FM is valid irrespective of other diagnoses. A diagnosis of FM does not exclude the presence of other clinically important illnesses
* PTSD Checklist-Stressor-Specific Version 1 re-experiencing (intrusion) symptom, 3 avoidance (numbing) symptoms, and 2 hyperarousal symptoms, each present at the level of moderate or higher during the past month, and if the total severity score is 50 or higher

Inclusion Criteria for Veterans living without FM:

* Age-matched to participant with FM

Exclusion Criteria:

Exclusion Criteria for Veterans living with FM:

* Neurological disorder
* Body mass index > 40
* Chronic kidney disease
* Severe cardiac condition (chronic heart failure, stenosis, history of cardiac arrest, defibrillator, angina)
* Ischemic heart disease
* 90 days of daily opioid use
* Beta-blocker
* Inability to consent for study participation (9) Significant cognitive impairment, defined as a known diagnosis of dementia (10) MRI contraindications (11) Pregnancy

Exclusion Criteria for Veterans living without FM:

* Active use of medications affecting pain responses
* Neurological disorder
* Body mass index > 40
* MRI contraindications
* Pregnancy

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Dispositional Trait Styles | Baseline to 12 weeks
  As a measurement of affect, participants will complete the Positive and Negative Affect Schedule and indicate the frequency with which the participants generally experience 10 positive (i.e., interested, excited) and 10 negative (i.e., distressed, upset) feelings. Items are rated ranging from 1 (very slightly or not at all) to 5 (extremely) with a total subscale ranging from 10 to 50.
Feasibility | Baseline to 12 weeks
  Feasibility will be percentage of exercise sessions attended.
Clinical Pain Severity | Baseline to 12 weeks
  Participants will self-report a number between 0-100 describing the intensity of pain, such that 0= no pain and 100 = the most intense pain imaginable. Any integer from 0 to 100 can be provided.
Pain Threshold | Baseline to 12 weeks
  Pain threshold refers to the intensity at which a stimulus is first perceived as painful. Pressure stimuli will be delivered to the participant's forearm and lower back using a handheld pressure algometer. The pressure will gradually increase until the participant responds by pressing a button on a handheld device. For pressure threshold, participants will be instructed to press the button when the sensation "first becomes painful."
Temporal Summation of Pain | Baseline to 12 weeks
  Temporal summation refers to a form of endogenous pain facilitation characterized by the perception of increased pain despite constant or even reduced peripheral afferent input. Temporal summation is presumed to be the psychosocial manifestation of wind-up. Wind-up is a phenomenon where repetitive stimulation of C primary afferents at rates greater that 0.3 Hertz produces a slowly increasing response of second-order neurons in the spinal cord. Temporal summation will be assessed using a nylon monofilament calibrated to bend a 300g of pressure on the back of the hand and lower back. Participants will be instructed to provide a verbal 0-100 rating of pain following a single contact of the monofilament. Then, participants will be instructed to provide another 0-100 rating of pain following a series of 10 contacts of the monofilament. This procedure will repeated twice at each location and pain ratings will be averaged across the two trials.
Conditioned Pain Modulation | Baseline to 12 weeks
  A routinely used quantitative sensory testing protocol for the measurement of endogenous pain inhibition is conditioned pain modulation, which refers to the reduction in pain from one stimulus (the test stimulus) produced by the application of a second pain stimulus at a remote body site (the conditioning stimulus). Conditioned pain modulation is believed to reflect the perceptual manifestation of diffuse noxious inhibitory controls, whereby ascending projections from one noxious stimulus activate supraspinal structures that trigger descending inhibitory projections to the dorsal horn. Participants will undergo four cold pressor immersions that consists of placing the non-dominant hand, up to the wrist, into circulating cold water for up to 1 minute and will provide a 0-100 rating of pain. Following each immersion, a handheld force algometer will be applied to either the forearm or lower back and press a handheld button to indicate when the pressure first becomes painful.
C-reactive protein | Baseline to 12 weeks
  A marker of pro-inflammation from blood draws
Tumor necrosis factor- alpha | Baseline to 12 weeks
  A marker of pro-inflammation from blood draws
Interleukin-6 | Baseline to 12 weeks
  A marker of pro-inflammation from blood draws
Interleukin- 10 | Baseline to 12 weeks
  A marker of pro-inflammation from blood draws
Interleukin- 8 | Baseline to 12 weeks
  A marker of pro-inflammation from blood draws
Myo-inositol | Baseline to 12 weeks
  marker of neuroinflammation measured via magnetic resonance spectroscopy imaging.
N-acetylaspartate | Baseline to 12 weeks
  marker of neuroinflammation measured via magnetic resonance spectroscopy imaging.
Choline | Baseline to 12 weeks
  marker of neuroinflammation measured via magnetic resonance spectroscopy imaging.
Lactate | Baseline to 12 weeks
  marker of neuroinflammation measured via magnetic resonance spectroscopy imaging.
Creatine | Baseline to 12 weeks
  marker of neuroinflammation measured via magnetic resonance spectroscopy imaging.
Brain Temperature | Baseline to 12 weeks
  marker of neuroinflammation using absolute brain temperatures (in °C) from magnetic resonance spectroscopy imaging.
Exercise Benefits and Barriers | Baseline to 12 weeks
  Participants will be asked to complete the Exercise Barriers and Benefits Scale that assesses perceived benefits and barriers to exercise to rank agreement with 29 statements, where 4='strongly agree' and 1='strongly disagree.'
Exercise Perceptions | Baseline to 12 weeks
  Semi-structured interviews will be conducted around topics related to current exercise behavior and any barriers the participants have to current exercise behavior, and will elicit participants' views on what an ideal exercise program would be.

CONTACTS AND LOCATIONS:
Overall Officials: Taylor L Taylor, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No